CLINICAL TRIAL: NCT00759070
Title: Effects of 2 Initial Standard Antiretroviral Combinations Therapies on Lipid Metabolism in ARV-naive HIV-infected Subjects
Brief Title: Effects of 2 Initial Standard Antiretroviral Combinations Therapies on Lipid Metabolism
Acronym: LIPOTAR-07
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juan A. Arnaiz (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, MD, PhD, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIPOTAR-07; EudraCT number: 2007-002698-29
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: Treatment Naïve
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; efavirenz; Lopinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tenofovir (TDF) + emtricitabine (FTC) + efavirenz (EFV)
  Interventions: Drug: Tenofovir + emtricitabine + efavirenz
- 2 (Active Comparator): Tenofovir (TDF) + emtricitabine (FTC) + lopinavir/ritonavir (LPV/RTV)
  Interventions: Drug: Tenofovir + emtricitabine + lopinavir/ritonavir

INTERVENTIONS:
Drug: Tenofovir + emtricitabine + efavirenz — Tenofovir 300 mg + emtricitabine 200 mg, (Truvada, Gilead Sciences)
  + Efavirenz 600 mg, (Sustiva, Bristol-Myers Squibb) once daily
  Arms: 1
Drug: Tenofovir + emtricitabine + lopinavir/ritonavir — Tenofovir 300 mg + emtricitabine 200 mg, (Truvada, Gilead Sciences)QD Lopinavir/ritonavir 400 mg/100 mg, (Kaletra, Abbott) BID
  Arms: 2

SUMMARY:
This study is an open-label, randomized, pilot comparison of the effects of either lopinavir/ritonavir or efavirenz in combination with tenofovir plus emtricitabine on cholesterol metabolism, mitochondrial functioning and immune response in 50 naive HIV patients after 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HIV-1 infection
* Age 18 or above
* Antiretroviral-naive
* Criteria for antiretroviral therapy in accordance with current guidelines
* Plasma LDL-cholesterol below 190 mg/dL
* Not receiving lipid-lowering agents
* Written informed consent

Exclusion Criteria:

* Use of phytosterol-enriched food previous month.
* Pregnancy or breastfeeding
* Cardiovascular disease
* Secondary Hypercholesterolemia
* Plasma creatinine above 1,2 mg/dL)
* Aminotransferases above 5 times ULN
* Current treatment for hepatitis C coinfection
* Diabetes mellitus (fasting glycemia > 124 mg/dL)
* Illegal drug use or alcohol abuse
* Active AIDS-defining opportunistic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Changes in total cholesterol and HDL and LDL fractions | 48 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Joan XXIII, Tarragona, Tarragona

REFERENCES:
- [Derived] Leyes P, Cofan M, Gonzalez-Cordon A, de Lazzari E, Trabal J, Domingo P, Negredo E, Vidal F, Forga MT, Gatell JM, Ros E, Martinez E. Increased cholesterol absorption rather than synthesis is involved in boosted protease inhibitor-associated hypercholesterolaemia. AIDS. 2018 Jun 19;32(10):1309-1316. doi: 10.1097/QAD.0000000000001837. PMID 29683854
- [Derived] Egana-Gorrono L, Martinez E, Domingo P, Lonca M, Escriba T, Fontdevila J, Vidal F, Negredo E, Gatell JM, Arnedo M. Differential subcutaneous adipose tissue gene expression patterns in a randomized clinical trial of efavirenz or lopinavir-ritonavir in antiretroviral-naive patients. Antimicrob Agents Chemother. 2014 Nov;58(11):6717-23. doi: 10.1128/AAC.03481-14. Epub 2014 Aug 25. PMID 25155608